## PHENOTYPING SEROCONVERSION FOLLOWING VACCINATION AGAINST COVID-19 IN PATIENTS ON HAEMODIALYSIS - SAP

**Sponsor Reference No: 0810** 

Date and Version No: 01.04.2021 Version 1

IRAS: 292716

Chief Investigator: Dr Matthew Graham-Brown – NIHR Academic Clinical Lecturer in

Renal medicine, Department of Cardiovascular Sciences, University of Leicester, and Honorary Specialist Registrar Renal Medicine, John Walls Renal Unit, University Hospitals Leicester.

Investigators: Professor Nigel Brunskill

Dr Richard Baines

**Professor James Burton** 

Dr Rupert Major

Dr Haresh Selvaskanden

Dr Katherine Hull

Miss Rosey Billany

Dr Sherna Adenwalla

Sponsor: University of Leicester

Funder: Leicester Charity Hospitals

Signatures: The approved protocol should be signed by author(s) and/or

person(s) authorised to sign the protocol

## **Confidentiality Statement**

All information contained within this protocol is regarded as, and must be kept confidential. No part of it may be disclosed by any Receiving Party to any Third Party, at any time, or in any form without the express written permission from the Chief Author/Investigator and / or Sponsor.

## Quantitative Analysis:

Statistical analyses will be performed using SPSS and GraphPad Prism. Descriptive data will be presented as mean +/- standard deviation and median [interquartile range] for normally and non-normally distributed data respectively. Exploratory analyses will be undertaken with Chi-squared and independent samples t-tests to look for potential patient-related factors which may account for differences in seroconversion.

The Number of Participants

This study will include 115 participants. 95 patients with ESKD on haemodialysis and 20 healthy volunteers

The Level of Statistical Significance  $\alpha$ = 0.05

Procedure for Accounting for Missing, Unused, and Spurious Data.

Missing data will be handled by imputation of last variable carried forward (assumption of no change).